CLINICAL TRIAL: NCT00187668
Title: Study Of PHarmacogenetics in Ethnically Diverse Populations (SOPHIE Study)
Acronym: SOPHIE
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 701
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Focus Groups
Keywords: Healthy Cohort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 40 mL of blood for DNA extraction
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- African American: Must self identify as African American with parents and grandparents of the same ethnicity. Must be healthy taking no over the counter medications or prescription medications.
- Cuacasian: Must self identify as Caucasian with parents and grandparents of the same ethnicity. Must be healthy taking no over the counter medications or prescription medications.
- Hispanic: Must self identify as Hispanic with parents and grandparents of the same ethnicity. Must be healthy taking no over the counter medications or prescription medications.
- Asian: Must self identify as Asian with parents and grandparents of the same ethnicity. Must be healthy taking no over the counter medications or prescription medications.

SUMMARY:
Collect DNA from well-characterized healthy volunteers.

DETAILED DESCRIPTION:
DNA and plasma will be used to identify and determine allele frequencies of genetic variants in membrane transporters and other genes relevant to human disease or drug response, including drug metabolizing enzymes, collagen, race/ethnicity, neurovascular disease, asthma/allergy/lung disease, and cardiovascular disease. This phase of the study will serve as the hypothesis-generating phase for future studies by identifying genetic variants and determining allele frequencies among an ethnically diverse cohort of healthy volunteers. Future investigations (separate IRB applications) will attempt to correlate genotypes to phenotypes among this cohort of volunteers. The allele identification and frequency data from this group of healthy volunteers will also be used to design association studies in relevant disease populations.

Determine if identified sequence variants are associated with gain or loss of in vitro biologic function using lymphocytes obtained from patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects of both genders and specified ethnic groups
* Subjects must be between 18-40 years of age

Exclusion Criteria:

* Smokers
* Drink > 2 alcoholic beverages/day
* Take any chronic medication

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy participants that are willing to be called back for subsequent genotype to phenotype studies.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2004-02; Primary Completion 2023-08 (Actual); Study Completion 2023-08 (Actual)

PRIMARY OUTCOMES:
Healthy Control | On-going
  Amass a cohort of healthy controls to be used for future genotype to phenotype studies.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Giacomini, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hopsital CTSI CRC, San Francisco, California, United States

REFERENCES:
- [Background] Ha Choi J, Wah Yee S, Kim MJ, Nguyen L, Ho Lee J, Kang JO, Hesselson S, Castro RA, Stryke D, Johns SJ, Kwok PY, Ferrin TE, Goo Lee M, Black BL, Ahituv N, Giacomini KM. Identification and characterization of novel polymorphisms in the basal promoter of the human transporter, MATE1. Pharmacogenet Genomics. 2009 Oct;19(10):770-80. doi: 10.1097/FPC.0b013e328330eeca. PMID 19745787
- [Background] Urban TJ, Sebro R, Hurowitz EH, Leabman MK, Badagnani I, Lagpacan LL, Risch N, Giacomini KM. Functional genomics of membrane transporters in human populations. Genome Res. 2006 Feb;16(2):223-30. doi: 10.1101/gr.4356206. Epub 2005 Dec 14. PMID 16354753
- [Background] Shu Y, Leabman MK, Feng B, Mangravite LM, Huang CC, Stryke D, Kawamoto M, Johns SJ, DeYoung J, Carlson E, Ferrin TE, Herskowitz I, Giacomini KM; Pharmacogenetics Of Membrane Transporters Investigators. Evolutionary conservation predicts function of variants of the human organic cation transporter, OCT1. Proc Natl Acad Sci U S A. 2003 May 13;100(10):5902-7. doi: 10.1073/pnas.0730858100. Epub 2003 Apr 28. PMID 12719534
- [Background] Kroetz DL, Pauli-Magnus C, Hodges LM, Huang CC, Kawamoto M, Johns SJ, Stryke D, Ferrin TE, DeYoung J, Taylor T, Carlson EJ, Herskowitz I, Giacomini KM, Clark AG; Pharmacogenetics of Membrane Transporters Investigators. Sequence diversity and haplotype structure in the human ABCB1 (MDR1, multidrug resistance transporter) gene. Pharmacogenetics. 2003 Aug;13(8):481-94. doi: 10.1097/00008571-200308000-00006. PMID 12893986
- [Background] Gray JH, Mangravite LM, Owen RP, Urban TJ, Chan W, Carlson EJ, Huang CC, Kawamoto M, Johns SJ, Stryke D, Ferrin TE, Giacomini KM. Functional and genetic diversity in the concentrative nucleoside transporter, CNT1, in human populations. Mol Pharmacol. 2004 Mar;65(3):512-9. doi: 10.1124/mol.65.3.512. PMID 14978229
- [Background] Badagnani I, Chan W, Castro RA, Brett CM, Huang CC, Stryke D, Kawamoto M, Johns SJ, Ferrin TE, Carlson EJ, Burchard EG, Giacomini KM. Functional analysis of genetic variants in the human concentrative nucleoside transporter 3 (CNT3; SLC28A3). Pharmacogenomics J. 2005;5(3):157-65. doi: 10.1038/sj.tpj.6500303. PMID 15738947
- [Background] Owen RP, Gray JH, Taylor TR, Carlson EJ, Huang CC, Kawamoto M, Johns SJ, Stryke D, Ferrin TE, Giacomini KM. Genetic analysis and functional characterization of polymorphisms in the human concentrative nucleoside transporter, CNT2. Pharmacogenet Genomics. 2005 Feb;15(2):83-90. doi: 10.1097/01213011-200502000-00004. PMID 15861032